CLINICAL TRIAL: NCT05539196
Title: A Post-Approval Registry for Exablate 4000 Type 1.0 and Type 1.1 for Unilateral Pallidotomy for the Treatment of Advanced, Idiopathic Parkinson's Disease With Medication-refractory Moderate to Severe Motor Complications
Status: Recruiting | Type: Observational
Sponsor: InSightec (Industry)
Responsible Party: Sponsor
Other Study IDs: PD006PAS/PD015
Record Dates: First submitted 2022-09-12; First posted 2022-09-14 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Movement Disorders; Neurology; Parkinsons Disease
MeSH Terms: conditions — Movement Disorders; Parkinson Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

GROUPS / COHORTS (1):
- Post Exablate Neuro Pallidotomy for Parkinson's Disease with Motor Complications: The population enrolled in this registry will be comprised of male and female patients that plan to be treated using the Exablate Neuro system for advanced, idiopathic Parkinson's disease with medication-refractory moderate to severe motor complications. No intervention is performed under this registry protocol.
  Interventions: Device: Exablate Pallidotomy, Unilateral

INTERVENTIONS:
Device: Exablate Pallidotomy, Unilateral — Unilateral pallidotomy using focused ultrasound for the treatment of Parkinson's Disease with medication-refractory moderate to severe motor complications.

SUMMARY:
This registry is a prospective, multicenter, international, single arm, observational post-approval registry with follow-up at 3, 6, and 12 months, and annually for 5 years. The proposed registry will enroll 60 subjects and will be conducted at approximately 10 centers worldwide.

DETAILED DESCRIPTION:
This is a post-approval registry which is required by of the approval under PMA P150038/S014 for the Exablate® Model 4000 (Exablate Neuro) Type 1.0 and Type 1.1 for unilateral pallidotomy in the treatment of idiopathic Parkinson's Disease with medication-refractory moderate to severe motor complications. Subjects participating in this registry will have received a unilateral pallidotomy using the commercially available Exablate Neuro.

The following assessments will be collected at Baseline, 3, 6, and 12 months post Exablate procedure and annually thereafter for 5 years:

Adverse Events (AEs) (does not apply to Baseline Visit) Medication usage MDS-UPDRS Unified Dyskinesia Rating Scale EQ-5D-5L WPAI-GH Clinician and Patient Global Impression of Change Patient Satisfaction Questionnaire

ELIGIBILITY:
Inclusion Criteria:

* Men and women, age 30 years and older.
* Subject undergoing a planned an Exablate procedure for their Parkinson's Disease with Motor Complications per local institution standard of care.
* Subject is willing to cooperate with the Registry requirements including compliance with the regimen and completion of all Registry visits.
* Subject has signed and received a copy of the approved informed consent form.

Exclusion Criteria:

* Subject does not agree to participate or is unlikely to participate for the entirety of the Registry.

Ages: 30 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The population enrolled in this registry will be comprised of male and female patients that plan to be treated using the Exablate Neuro system for advanced, idiopathic Parkinson's disease with medication-refractory moderate to severe motor complications. Subjects must meet the specific eligibility criteria in order to enroll in this Registry.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2023-01-23 (Actual); Primary Completion 2029-07-31 (Estimated); Study Completion 2029-07-31 (Estimated)

PRIMARY OUTCOMES:
Responder Analysis | 5 years
  Primary Effectiveness will be evaluated through a Responder analysis. Responder is defined as the patient reaching a minimally clinically significant difference on: 1) UDysRS Objective Assessment ON Meds, without clinically significant worsening of MDS-UPDRS Part III OFF Meds aggregated extremity score for treated side Or 2) MDS-UPDRS Part III OFF Meds Motor Exam on the treated side, without clinically significant worsening of UDysRS Objective Assessment ON meds

OTHER OUTCOMES:
Safety Analysis | 5 years
  Safety will be evaluated through descriptive analysis of the incidence and severity of adverse events. Adverse events will be recorded and categorized according to severity, expectedness, and relationship to Exablate Neuro system pallidotomy procedure and/or disease progression.

CONTACTS AND LOCATIONS:
Locations (5):
- United States (4):
  - University of Maryland, Baltimore, Baltimore, Maryland
  - Weill Cornell Medicine, New York, New York
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - University of Texas Southwestern Medical Center, Dallas, Texas
- Ohnishi Neurological Center, Akashi, Hyōgo, Japan